CLINICAL TRIAL: NCT01755923
Title: A Phase Ⅱ Randomized Controlled Trial to Compare Gefitinib With Docetaxel as Second-line Therapy for Advanced or Metastatic Non-squamous NSCLC Patients With Wild-type EGFR
Brief Title: Gefitinib or Docetaxel as Second Line Therapy for Wild-type Epidermal Growth Factor Receptor (EGFR) NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-S466
Record Dates: First submitted 2012-12-17; First posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; wild-type EGFR; gefitinib; docetaxel; second-line therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gefitinib (Experimental): Gefitinib (Iressa) 250mg once per day until progression disease or intolerant side effects
  Interventions: Drug: Gefitinib
- Docetaxel (Active Comparator): Docetaxel 75mg/m2,d1,every 3 weeks, at least 2-6 cycles depending on the progression disease or the patient's physical condition
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250mg once per day until the progression disease or intolerant side effects
  Other Names: Iressa
  Arms: Gefitinib
Drug: Docetaxel — Docetaxel 75mg/m2 iv, d1,every 3 weeks, at least 2-6 cycles depending on the progression disease or the patient's physical condition
  Other Names: Taxotere
  Arms: Docetaxel

SUMMARY:
Gefitinib, the first EGFR-tyrosine kinase inhibitor (TKI) in the world was examined as monotherapy in two phase Ⅱ studies called IDEAL trials. Response rate with doses of 250mg and 500mg/day were similar, ranging from 10% to 18%. Posterior analysis demonstrated that patients with EGFR mutation had an improved response rate (RR) to gefitinib compared to wild-type patients (46% versus 10%). The early trials that evaluated EGFR-TKIs for the second- and third-line settings of advanced NSCLC did not select patients on the basis of any EGFR marker. The IEESSA Survival Evaluation in Lung Cancer (ISEL) trial evaluated the role of second-line gefitinib 250mg/day in 1692 patients with advanced NSCLC. Patients with EGFR mutations had higher RR than patients without (37.5% versus 2.6%). From the above results, the response rate in patients without EGFR gene mutation was obviously different (10% versus 2.6%). The methods used for detecting EGFR gene mutation was different, which might contribute to the difference of response rates. In IDEAL trial, EGFR gene mutation was detected by sequencing. But in ISEL trial, EGFR gene mutation was detected by ARMS. As we know, ARMS was more sensitive than sequencing in detecting EGFR gene mutation. That is to say, in IDEAL trials some EGFR mutant patients were misdiagnosed as wild-type patients, so the response rate was higher. Recently, Wu Yi-Long et al reported that relative abundance of EGFR mutations predicted benefit form gefitinib treatment for advanced non small cell lung cancer. The study cohort was all Chinese. In this study, the objective response rate in patients without EGFR mutation detected by ARMS was 16.1%, which was significantly higher than the response rate of docetaxel. But in 2012 American society of clinical oncology (ASCO) annual meeting, the Tailor study in which Italian NSCLC patients were enrolled demonstrated a clear superiority of docetaxel over erlotinib as second line treatment for patients without EGFR mutations in exons 19 or 21. So we wonder if the racial difference is the determinant factor. So the purpose of this trial is to compare the efficacy and safety of gefitinib with docetaxel as second-line therapy for advanced or metastatic Chinese NSCLC patients with wild-type EGFR.

DETAILED DESCRIPTION:
The adoption of docetaxel as a standard second line therapy was based on data from two phase Ⅲ trials. In the first trail, docetaxel (75mg/m2, every 3 weeks) significantly prolonged median and 1-year survival duration compared with best supportive care (median survival, 7.5 months versus 4.6 months; P=0.010; 1-year survival, 37% versus 12%), although the response rate was low (5.5%). In the second study the 6-months and median survival rates were similar for docetaxel and vinorelbine or ifosfamide. However, the 1-year survival rate was significantly greater with docetaxel than ifosfamide or vinorelbine (32% versus 19%, P=0.025). In both studies docetaxel significantly improved some parameters of quality of life. Since these two pivotal studies, new potential second-line drugs were compared with the docetaxel standard of care. With regards to the therapeutic results of the docetaxel arm of these studies, it must be emphasized that response rates and survival data were highly and significantly reproducible.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Life expectancy more than 12 weeks
* histologically or cytologically confirmed inoperable non-squamous NSCLC (stage ⅢB/Ⅳ)
* ineligible for curative radiotherapy
* no prior radiotherapy for the target lesions
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* previous treatment include first-line platinum doublet chemotherapy
* no EGFR gene mutation detected by Scorpions-ARMS
* at least one bidimensionally measurable or radiographically assessable lesion
* adequate bone marrow reserve
* adequate hepatic and renal function

Exclusion Criteria:

* prior treatments including any of the following drugs: gefitinib and docetaxel
* additional malignancies
* uncontrolled systemic disease
* any evidence of clinically active interstitial lung disease
* newly diagnosed central nervous system (CNS)metastasis and not treated by radiotherapy of surgery
* pregnancy or breast feeding phase

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 52 weeks (about one year)
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks.

SECONDARY OUTCOMES:
Overall survival | Up to 100 weeks
  From the date of randomization until the date of death from any cause, assessed up to 100 weeks.
Objective response rate | up to 9 weeks
  The objective response rate includes the complete remission and partial remission rate.
the score of functional assessment of cancer treatment-lung (FACT-L) | up to 100 weeks
  FACT-L is assessed at different time points.(Date of randomization, 1 week after chemotherapy/EGFR-TKI, every cycle of chemotherapy/EGFR-TKI, every month of EGFR-TKI treatment/observation, up to 100 weeks)
Number of participants with adverse events | Up to 6 months
  The adverse events are assessed by National Cancer Institute-Common Toxcity Criteria (Version 3.0)(NCI-CTC).

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Respiratory Medicine, Peking Union Medical College Hospita, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Shepherd FA, Dancey J, Ramlau R, Mattson K, Gralla R, O'Rourke M, Levitan N, Gressot L, Vincent M, Burkes R, Coughlin S, Kim Y, Berille J. Prospective randomized trial of docetaxel versus best supportive care in patients with non-small-cell lung cancer previously treated with platinum-based chemotherapy. J Clin Oncol. 2000 May;18(10):2095-103. doi: 10.1200/JCO.2000.18.10.2095. PMID 10811675
- [Result] Fossella FV, DeVore R, Kerr RN, Crawford J, Natale RR, Dunphy F, Kalman L, Miller V, Lee JS, Moore M, Gandara D, Karp D, Vokes E, Kris M, Kim Y, Gamza F, Hammershaimb L. Randomized phase III trial of docetaxel versus vinorelbine or ifosfamide in patients with advanced non-small-cell lung cancer previously treated with platinum-containing chemotherapy regimens. The TAX 320 Non-Small Cell Lung Cancer Study Group. J Clin Oncol. 2000 Jun;18(12):2354-62. doi: 10.1200/JCO.2000.18.12.2354. PMID 10856094
- [Result] Hanna N, Shepherd FA, Fossella FV, Pereira JR, De Marinis F, von Pawel J, Gatzemeier U, Tsao TC, Pless M, Muller T, Lim HL, Desch C, Szondy K, Gervais R, Shaharyar, Manegold C, Paul S, Paoletti P, Einhorn L, Bunn PA Jr. Randomized phase III trial of pemetrexed versus docetaxel in patients with non-small-cell lung cancer previously treated with chemotherapy. J Clin Oncol. 2004 May 1;22(9):1589-97. doi: 10.1200/JCO.2004.08.163. PMID 15117980
- [Result] Cufer T, Vrdoljak E, Gaafar R, Erensoy I, Pemberton K; SIGN Study Group. Phase II, open-label, randomized study (SIGN) of single-agent gefitinib (IRESSA) or docetaxel as second-line therapy in patients with advanced (stage IIIb or IV) non-small-cell lung cancer. Anticancer Drugs. 2006 Apr;17(4):401-9. doi: 10.1097/01.cad.0000203381.99490.ab. PMID 16549997
- [Result] Fukuoka M, Yano S, Giaccone G, Tamura T, Nakagawa K, Douillard JY, Nishiwaki Y, Vansteenkiste J, Kudoh S, Rischin D, Eek R, Horai T, Noda K, Takata I, Smit E, Averbuch S, Macleod A, Feyereislova A, Dong RP, Baselga J. Multi-institutional randomized phase II trial of gefitinib for previously treated patients with advanced non-small-cell lung cancer (The IDEAL 1 Trial) [corrected]. J Clin Oncol. 2003 Jun 15;21(12):2237-46. doi: 10.1200/JCO.2003.10.038. Epub 2003 May 14. PMID 12748244
- [Result] Kris MG, Natale RB, Herbst RS, Lynch TJ Jr, Prager D, Belani CP, Schiller JH, Kelly K, Spiridonidis H, Sandler A, Albain KS, Cella D, Wolf MK, Averbuch SD, Ochs JJ, Kay AC. Efficacy of gefitinib, an inhibitor of the epidermal growth factor receptor tyrosine kinase, in symptomatic patients with non-small cell lung cancer: a randomized trial. JAMA. 2003 Oct 22;290(16):2149-58. doi: 10.1001/jama.290.16.2149. PMID 14570950
- [Result] Bell DW, Lynch TJ, Haserlat SM, Harris PL, Okimoto RA, Brannigan BW, Sgroi DC, Muir B, Riemenschneider MJ, Iacona RB, Krebs AD, Johnson DH, Giaccone G, Herbst RS, Manegold C, Fukuoka M, Kris MG, Baselga J, Ochs JS, Haber DA. Epidermal growth factor receptor mutations and gene amplification in non-small-cell lung cancer: molecular analysis of the IDEAL/INTACT gefitinib trials. J Clin Oncol. 2005 Nov 1;23(31):8081-92. doi: 10.1200/JCO.2005.02.7078. Epub 2005 Oct 3. PMID 16204011
- [Result] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Result] Thatcher N, Chang A, Parikh P, Rodrigues Pereira J, Ciuleanu T, von Pawel J, Thongprasert S, Tan EH, Pemberton K, Archer V, Carroll K. Gefitinib plus best supportive care in previously treated patients with refractory advanced non-small-cell lung cancer: results from a randomised, placebo-controlled, multicentre study (Iressa Survival Evaluation in Lung Cancer). Lancet. 2005 Oct 29-Nov 4;366(9496):1527-37. doi: 10.1016/S0140-6736(05)67625-8. PMID 16257339
- [Result] Hirsch FR, Varella-Garcia M, Bunn PA Jr, Franklin WA, Dziadziuszko R, Thatcher N, Chang A, Parikh P, Pereira JR, Ciuleanu T, von Pawel J, Watkins C, Flannery A, Ellison G, Donald E, Knight L, Parums D, Botwood N, Holloway B. Molecular predictors of outcome with gefitinib in a phase III placebo-controlled study in advanced non-small-cell lung cancer. J Clin Oncol. 2006 Nov 1;24(31):5034-42. doi: 10.1200/JCO.2006.06.3958. PMID 17075123